CLINICAL TRIAL: NCT01220089
Title: Adaptation of the Diabetes Prevention Program for Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0719; K24DK065018 (NIH); 10SDG210292 (Other)
Record Dates: First submitted 2010-09-23; First posted 2010-10-13 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: obesity; weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard maintenance (Active Comparator): During months 7 to 18, individuals in the Standard Maintenance condition will receive informational handouts by mail (or e-mail) regarding weight maintenance.
  Interventions: Behavioral: Standard maintenance
- Intensified Maintenance (Active Comparator): During months 7 to 18, individuals in the Intensified Maintenance condition will continue to have monthly in-person visits with the weight loss counselor ("Weight Coach").
  Interventions: Behavioral: Intensified maintenance

INTERVENTIONS:
Behavioral: Standard maintenance — Participants will receive written materials in months 7-18
  Arms: Standard maintenance
Behavioral: Intensified maintenance — Participants will continue with in-person counseling visits in months 7-18
  Arms: Intensified Maintenance

SUMMARY:
The study has two primary aims. The first aim is to assess the efficacy of adding in-person visits to the use of portion-controlled foods for long-term weight loss. The second aim is to assess the use of trained lay counselors for the maintenance of weight loss. The primary endpoint of the study will be changes in weight. Secondary endpoints will include changes in body mass index (BMI), cardiovascular risk factors, health-related quality of life, and cost-effectiveness. The addition of in-person visits with the weight loss counselor is predicted to lead to greater long-term weight loss than the use of portion-controlled foods alone.

DETAILED DESCRIPTION:
This study will be a randomized trial of a weight control intervention, with participants recruited primarily from primary care practices at the University of Colorado. Study treatment will be delivered at the Center for Human Nutrition, an inter-disciplinary research clinic which is part of the University of Colorado School of Medicine. If needed, administrative study visits, such as for informed consent and for completion of questionnaires, may take place at offices in the Division of General Internal Medicine. Up to 200 patients will be enrolled, of which up to 125 will be provided with 6 months of high-intensity weight loss counseling. During the first 6 months, each participant will be seen for 12 counseling visits. These visits will take place at weeks 1, 2, 3, 4, 6, 8, 10, 12, 15, 18, 21, and 24. We estimate that between 10% and 20% of these patients will drop out prior to 6 months. After the first 6 months, the remaining participants will be randomly assigned to a treatment condition: Standard Maintenance or Intensified Maintenance. During months 7 to 18, individuals in the Standard Maintenance condition will receive informational handouts by mail (or e-mail) regarding weight maintenance, while those in the Intensified Maintenance condition will continue to have monthly in-person visits with the weight loss counselor ("Weight Coach").

All participants will use portion-controlled foods to replace 2 meals per day during the first 6 months of treatment and to replace 1 meal per day during months 7 to 18. Participants will purchase their own portion-controlled foods, although in-kind contributions from private industry will be sought to offset participants' food costs. The study consent form will explicitly describe estimated food costs for study participants. The cost of the meal plan, a "partial meal replacement" diet (replacement of 2 out of 3 meals per day) is not expected to increase food costs. Many participants should observe a decrease in food costs while following the meal plan.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 79
* Able to give informed consent
* Able to keep a food record for 7 days prior to study entry and to complete 2 screening visits and a blood draw prior to enrollment
* Willing to attend all counseling sessions, to complete study-related assessments, and to be randomized to a treatment condition after 6 months of treatment
* Has a regular primary care physician (if referred from outside the University of Colorado system)
* Body mass index (BMI) ≥ 30 kg/m2 and < 50 kg/m2
* Elevated waist circumference (≥ 88 cm for women, ≥ 102 cm for men) + any one of the following:
* Glucose intolerance (fasting glucose ≥ 100 or non-fasting glucose ≥ 140, including type 2 diabetes); individuals taking medications for diabetes qualify automatically
* Elevated blood pressure (≥ 130/85), including hypertension (≥ 140/90); individuals taking anti-hypertensive medication qualify automatically
* Hyperlipidemia/dyslipidemia, including any of the following: hypertriglyceridemia (TG ≥ 150); low HDL cholesterol (< 40 for men, < 50 for women); or taking lipid-lowering medications
* Obstructive sleep apnea -

Exclusion Criteria:

* Medical conditions in which significant weight loss is normally contraindicated (e.g. pregnancy, congestive heart failure requiring diuretics, poorly controlled diabetes, Stage 4 or 5 chronic kidney disease, clinically evident cirrhosis, other severe internal organ disease); exceptions may be made if a referring physician documents that it is safe and appropriate for the individual to lose weight
* Treated for cancer within the past 5 years, except for basal cell or squamous cell skin cancer; exceptions may be made with written permission from a physician
* Myocardial infarction or stroke within the past 6 months
* Poorly controlled hypertension (≥ 160/100); may be re-screened when controlled
* Poorly controlled diabetes (hemoglobin A1c ≥ 10.0); may be re-screened when controlled
* Weight gain or loss of ≥ 5% of weight in the past 6 months; patients who have not been weight stable may be re-screened
* Chronic use of corticosteroids or second-generation antipsychotic medications (exceptions may be made for individuals using these medications who have been weight stable for 6 months)
* Psychiatric diagnoses likely to affect adherence to a research study protocol (e.g., poorly controlled schizophrenia, active substance abuse)
* Untreated major depression (PHQ-9 score ≥ 20)
* Pregnant or trying to become pregnant
* Social situation precluding participation in a research study (e.g., need to care for a small child or an elderly parent)
* Prior or planned bariatric surgery
* Participation in an organized weight loss program (e.g., Weight Watchers) at the time of enrollment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
weight change | Weeks 1-4, 6, 8, 10, 12, 15, 18, 21, 24 & 72

SECONDARY OUTCOMES:
change in glucose | baseline, 6 months & 18 months
change in blood pressure | baseline, 6 months & 18 months
change in waist circumference | baseline, 6 months & 18 months
change in lipids | baseline, 6 months & 18 months
change in health-related quality of life | baseline & 18 months
cost effectiveness | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam G Tsai, MD, MSCE, Principal Investigator — University of Colorado, Denver
Locations (1):
- Center for Human Nutrition, Denver, Colorado, United States

REFERENCES:
- [Derived] Tsai AG, Juarez-Colunga E, Felton S, Speer RB, Bessesen DH, Atherly AJ. Medication costs during an 18 month clinical trial of obesity treatment among patients encountered in primary care. BMC Obes. 2015 May 29;2:24. doi: 10.1186/s40608-015-0054-4. eCollection 2015. PMID 26217539